CLINICAL TRIAL: NCT04415385
Title: The Combination of Camrelizumab and Apatinib as Second-line Therapy for Advanced Pancreatic Cancer Patients Who Failed Standard First-line Treatment: a Single Arm, Open-label, Phase 2 Study
Brief Title: The Combination of Camrelizumab and Apatinib as Second-line Therapy for Advanced Pancreatic Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChiECRCT20200088
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab + Apatinib (Experimental): Participants receive Camrelizumab 200mg intravenously every 2 weeks and apatinib 250mg orally once daily until disease progression or unacceptable toxicity
  Interventions: Drug: Camrelizumab; Drug: Apatinib

INTERVENTIONS:
Drug: Camrelizumab — 200mg, intravenous infusion for 30 minutes (including the time of the tube, the overall infusion time is not shorter than 20 minutes, no longer than 60 minutes), once every 2 weeks.
  Other Names: SHR-1210
Drug: Apatinib — 250 mg, orally once a day. Take about half an hour after a meal with warm water.
  Other Names: Apatinib Mesylate

SUMMARY:
This is an single arm, open-label, phase II trial to evaluate safety and efficacy of using the combination of Camrelizumab with apatinib as second-line therapy for advanced PDAC.

DETAILED DESCRIPTION:
PD-1 antibody Camrelizumab is a humanized monoclonal antibody, and the heavy chain is immunoglobulin G4 (IgG4), the light chain is immunoglobulin κ (IgK). Camrelizumab specifically binds to PD-1 and blocks the interaction of PD-1 with its ligand (PD-L1), allowing T cells to recover against tumor immune responses.

Response rate, progression-free survival, overall survival, duration of response，disease control rate, drugs related side effects were recorded and analyzed, to assess the combination treatment could or couldn't benefit the patients with advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily joined the study and signed informed consent. Able to comply with the required protocol and follow-up procedures;
2. Histologically or cytologically confirmed recurrent / metastatic advanced pancreatic cancer, have received gemcitabine or nab-paclitaxel based standard chemotherapy;
3. Male and Female, Age ≥ 18 years and ≤ 70 years;
4. Life expectancy exceeds 3 months;
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2;
6. Patients must have measurable disease per RECIST 1.1;
7. Subjects with previous systemic therapy completed more than 2 weeks can be enrolled,and the treatment-related AE should be restored to NCI-CTCAE v5.0 less than grade 1 (except for grade 2 hair loss)
8. Subjects with asymptomatic central nervous system metastasis, or asymptomatic brain metastases after treatment, need to be examined by CT or MRI, disease stable for at least 3 months, and at least 4 weeks without steroid medication;
9. Subjects must provide tumor tissue and blood samples for specific index testing;
10. The HBsAg test is negative; if the HBsAg or HBcAb test is positive, the HBV DNA test must be less than 1000 IU / ml;
11. The HCV-Ab test is negative; if the HCV-Ab or HCV-RNA test is positive, ALT and AST CTCAE v5 ≤ 1 level and ≤ 3 × ULN; The joint infection of hepatitis B and C shouled be excluded;
12. Subjects must have adequate organ function (without blood transfusion, without growth factor or blood components support within 14 days before enrollment)as determined by: Hemoglobin ≥ 9 g/dL; Absolute neutrophil count (ANC) ≥1.5×109/L; Platelet count ≥ 90×109/L ; Total bilirubin ≤ 1×upper limit of normal(ULN)；alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3×upper limit of normal(ULN), for subjects with liver metastases, ALT and AST≤5×ULN; Alkaline phosphatase ≤ 2.5 × upper limit of normal(ULN); urea nitrogen (BUN) and creatinine (Cr) ≤ 1.5 × upper limit of normal(ULN);
13. Women of childbearing age should agree to use contraceptives (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months of the end of the study; the serum or urine pregnancy test is negative within 7 days prior to study enrollment, and Must be non-lactating; males should agree to use contraceptives during the study period and within 6 months of the end of the study period.

Exclusion Criteria:

1. There is a third space effusion that cannot be controlled by drainage or other methods (e.g., large amounts of pleural and ascites), and the efficacy of clinical treatment cannot be evaluated;
2. Subjects who are ready to undergo or have previously undergone organ or bone marrow transplantation;
3. Subjects with known active CNS metastases or cancerous meningitis；
4. Surgical and/or radiotherapy failed to radically treated spinal cord compression, or previously diagnosed spinal cord compression did not have clinical evidence for disease stable more than 1 week before the first administration；
5. Imaging examination showed that there was a clear manifestation of tumor invading the abdominal great vessels；
6. Subjects with grade II or above myocardial ischemia, myocardial infarction, unstable angina pectoris and uncontrolled arrhythmia within six months before the first administration;
7. Subjects with grade III or IV cardiac insufficiency according to the New York Heart Association (NYHA) criteria or color Doppler chocardiography showed left ventricular ejection fraction (LVEF < 50%) ;
8. Peripheral neuropathy with CTCAE V5 ≥ grade II;
9. Human immunodeficiency virus (HIV) infection;
10. Subjects have active pulmonary tuberculosis;
11. Previous or current interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severe impairment of lung function, etc. may interfere with the detection and management of suspected drug-related pulmonary toxicity；
12. Subjects had known active or suspected autoimmune disease.Enrollment was allowed to be stable and did not require systemic immunosuppressive therapy；
13. Subjects received the vaccine within 28 days before the first use of the study drug；
14. Subjects requiring systemic corticosteroids (>10 mg/day prednisone or equivalent doses of the same drug) or other immunosuppressive therapy within 14 days before or during the first dose of the study drug.Enrollment was allowed if inhaled or topical steroids or adrenaline replacement therapy at a dose of <10 mg/day prednisone were allowed in the absence of active autoimmune disease；
15. Any active infection requiring systemic anti-infective treatment occurred within 14 days prior to the first administration of the study drug；
16. Radiotherapy, chemotherapy, surgical treatment or other targeted therapy for pancreatic cancer had been received within 1 week before the first administration of the study drug and had not progressed from previous treatment;
17. Major surgery was performed within 28 days before the first administration. The definition of major surgery in this study is that recovery time of at least 3 weeks after surgery is required to be able to accept the surgery treated in this study.Tumor aspiration or lymph node biopsy allowed enrollment；
18. Subjects received radical radiotherapy within 3 months before the first administration of the study drug;
19. Other anti tumor treatments may be received during the study interval.Such as chemotherapy or radiotherapy (except palliative radiotherapy);
20. Subjects have previously received anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137 or anti-CTLA-4 antibody treatment, or any other antibody or T cell co-stimulation drugs or any drugs that target immune checkpoint;
21. Participating in other clinical studies or planning to start this study is less than 14 days from the end of treatment in a previous clinical study;
22. Severe allergy to any monoclonal antibody or study drug excipient;
23. Women who are pregnant or breastfeeding, those with fertility who are unwilling or unable to take effective contraception;
24. Known history of psychotropic drug abuse or drug use. Subjects who have stopped drinking can be enrolled；
25. The investigator judged that the subjects had other factors that could lead to the forced termination of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
ORR | Through study completion, an average of 2 years.
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1

SECONDARY OUTCOMES:
PFS | Through study completion, an average of 2 years.
  Progression-free survival is defined as the duration from date of enrollment to the first occurrence of progression of disease or death from any cause
OS | Through study completion, an average of 2 years.
  Overall survival is defined as the duration from date of enrollment to the date of death from any cause.
DoR | Through study completion, an average of 2 years.
  DOR is defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first.
DCR | Through study completion, an average of 2 years.
  DCR is defined as the percentage of participants in the analysis population who have a CR, PR or stable disease (SD) per RECIST 1.1.
Incidence of Adverse Events (AEs) in the treatment of Camrelizumab in combination with apatinib | Through study completion, an average of 2 years.
  Number of participants with adverse events occurring up to 30 days after the last administration are evaluated and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No